CLINICAL TRIAL: NCT05522725
Title: The Use of Clinell Universal Wipes, Clinell Sporicidal Wipes, and Clinell EvaluClean Fluorescent Marker System, in Reducing Environmental Contamination and Acquisitions of Multidrug Resistant Organisms and Hospital Acquired Infections
Brief Title: The Impact of Bedside Wipes in Multi-patient Rooms: a Prospective, Crossover Trial Evaluating Infections and Survival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Gama Healthcare Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Purpose: Prevention
Other Study IDs: 124-16-ASF
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Hospital Acquired Infection
Keywords: Hospital Environment; MDRO; Multidrug resistant; Nosocomial infections; Cleaning Practices; High-touch surfaces; HAI
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: We conducted a clustered crossover trial at Shamir medical center from October 20, 2016 to January 19, 2018. Clusters were randomly assigned to use either single-use quaternary ammonium-based wipes (Clinell®; Watford, UK) or standard practices (reusable cloths, buckets and bleach (hypochlorite 1,000-5,000 ppm)) for cleaning of high-touch surfaces. Six-month intervention periods were implemented in alternating sequence, separated by a 4-week washout period. Five high-touch surfaces were monitored by fluorescent markers (EvaluClean®; Watford, UK), and for the presence of MDRO. Study outcomes were compared between periods using generalized estimating equations, Poisson regression and Cox proportional hazards models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention phase (Experimental): Single-use wipes installed at the bedside
  Interventions: Other: Single-use wipes installed at the bedside
- Non-intervention phase (No Intervention): Standard practice according to Israeli ministry of health (MOH)

INTERVENTIONS:
Other: Single-use wipes installed at the bedside
  Arms: Intervention phase

SUMMARY:
Multidrug resistant organisms (MDRO) are prevalent in hospitals and are associated with hospital-acquired infections (HAI). High-touch surfaces serve as reservoirs and fomites for MDRO transmission. The investigators quantified the impact of hanging single-use cleaning/disinfecting wipes in patients' immediate environment within multi-patient rooms. Pre-specified outcomes were: 1) HAI rate, 2) cleaning frequency, 3) MDRO room contamination, 4) new MDRO acquisitions, and 5) in-hospital mortality.

DETAILED DESCRIPTION:
The study will be conducted over 15 months; each study phase will last 6 months, with a pre-study period (1 month), a washout period (1 month) and a post study period (1 month).

1. Pre-study period: all rooms will be cleaned daily according to "common practice" which consists of using hypochlorite in a concentration of 1000 ppm (bleach) and reused cloths. The immediate environment (i.e., the 'patient's unit') of those with C. difficile carriage will be cleaned daily with hypochlorite 2000 ppm and upon discharge with hypochlorite 5000 ppm. This is the current "common practice" at AHMC.
2. Phase I: medicine A and B: high touch surfaces (e.g., bedrail, bedside tables, monitor, and cables) will be cleaned with Clinell® Universal Wipes, and the patient's unit of C. difficile carriers will be cleaned with Clinell® Sporicidal Wipes. The floor, walls, and sink, will still be cleaned with bleach. Medicine C and D: all rooms will be cleaned daily according to "common practice" as mentioned above.
3. Washout period in all Medicine departments A, B, C and D: all rooms will be cleaned daily according to "common practice" as mentioned above.
4. Phase II: medicine A and B: all rooms will be cleaned daily according to "common practice" as mentioned above. Medicine C and D: high touch surfaces (bedrail, bedside tables, monitor, cables) will be cleaned with Clinell® Universal Wipes, and the patient's unit of C. difficile carriers will be cleaned with Clinell® Sporicidal Wipes. The floor, walls, and sink, will still be cleaned with bleach.
5. Post-study period: all rooms will be cleaned daily according to "common practice" as mentioned above.

During the intervention phase, the whole department will be subjected to the intervention, regardless of the number of MDRO carriers present on the department (i.e. signifying the "colonization pressure" at the department). "Colonization pressure" will be continuously captured and recorded for future analyses.

All departments will perform, per local Infection Control regulations, rectal surveillance cultures upon admission to the department, to diagnose VRE, CRE-CP, and CRE-non-CP from certain populations: 1) patients directly transferred from another hospital; 2) patients directly transferred from another department inside AHMC; 3) functionally dependent patients (per Katz criteria); 4) residents of long-term care facilities; 5) patients who were hospitalized in an acute care hospital in the past six months; and 6) prisoners. In addition, every department selects one day per week for screening (rectally again) of 10 additional patients who are already hospitalized, but belong to high risk population for VRE and/or CRE colonization. In addition, once a week, a sputum screening culture for the presence of A. baumannii is obtained from all mechanically ventilated patients. No other surveillance cultures are performed in those Medicine departments, except theoretically as part of an outbreak investigation. The median departmental occupancy of all participating departments is 45 patients (the median number of mechanically ventilated patients in each department is 5). The patients' mix in all participating departments is equal, and patients are hospitalized in a certain department randomly. The departments are equal in structure, in the number of patients, and in its patients' characteristics.

All the surveillance for HAI determination and MDRO acquisitions are conducted routinely and continuously by the Infection Control team at AHMC. The primary investigator of this proposal serves as the head of Infection Control service and therefore is personally involved in the surveillances processes for those endpoints.

Frequency of cleaning will be assessed by Clinell® EvaluClean™ fluorescent marker system twice a week, on Mondays and Thursdays morning until afternoon, in all participating departments throughout the study period. The assessment will include the marking of five locations at a patient unit from each participating department, and the examination of the marks 4 hours later. The five location points are: 1) right bedrail, 2) the tray of the bedside table, 3) the binder that contains the fluid balance pages, hanging at the foot of the bed, 4) Strip for delivery and storage at the headboard of each bed, and 5) the bed itself.

Since the 4 study units are all identical in structure (in terms of room numbers and bed numbers), the patient units that will be randomly selected every week will be compatible. For example, in the first week, the patient units that could be randomly selected will be bed number 2 in room number 9 and bed number 1 in room number 2, in all 4-study units.

Clinical cultures are all processed at the AHMC clinical microbiology laboratory. No additional cultures will be obtained specifically for this protocol.

1. MRSA, VRE, A. baumannii, and P. aeruginosa will be determined according to a Vitek-2 automated system and according to CLSI breakpoints and criteria.
2. CRE-CP and CRE non-CP will be determined according to the Israeli MOH national diagnostic guidelines (2013) and based, again, on CLSI criteria.
3. Toxin-producing C. difficile will be determined based of a GDH-based serology test (C. DIFF QUIK CHEK COMPLETE®; Alere™) and if necessary (i.e., inconclusive serology test result: positive for C. difficile GDH antigen but negative for C. difficile toxins), will be confirmed by a PCR-based test (Xpert® C. difficile; Cepheid©). Samples will be processed according to national Israeli guidelines (2013) and according to CLSI criteria.
4. All MDROs will be stored in -700C for future molecular analyses

Representative MDROs will be typed later on for future detailed transmission dynamics investigations.

The laboratory will be blinded to the source of the cultures (i.e., the study department and study phase).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at one of four Medicine departments at Assaf Harofeh Medical Center: Medicine A, Medicine B, Medicine C, or Medicine D.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7725 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Device-related HAI rates | 12 months
  Central line associated bloodstream infections (CLABSI) and catheter-associated urinary tract infections (CAUTI), monitored in accordance to CDC criteria

SECONDARY OUTCOMES:
Frequency of cleaning | 12 months
  Invisible fluorescent marks at the patient unit will be examined to assess whether the location has been cleaned or not, using Clinell® EvaluClean™ fluorescent marker system. The endpoint would be presented as percents of adherence (i.e., the number of locations cleaned, divided by the overall number of locations what were marked).
MDRO environmental contamination | 12 months
  Environmental contamination measurements of MDRO were performed for all patients with a current or recent (prior two years) culture of MRSA, VRE, CRE, A. baumannii, or P. aeruginosa.
New MDRO acquisitions | 12 months
  MDRO included methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Enterococcus (VRE), carbapenemase-producing and non-carbapenemase-producing carbapenem-resistant Enterobacterales (CRE-CP and CRE-non-CP, respectively), and non-lactose fermenting Gram-negative bacilli (Acinetobacter baumannii, Pseudomonas aeruginosa)
In-hospital mortality | 12 months
  In-hospital mortality was collected from medical charts. The endpoint is defined as the proportion of patients with in-hospital deaths during the measurement period.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Marchaim, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weber DJ, Rutala WA, Miller MB, Huslage K, Sickbert-Bennett E. Role of hospital surfaces in the transmission of emerging health care-associated pathogens: norovirus, Clostridium difficile, and Acinetobacter species. Am J Infect Control. 2010 Jun;38(5 Suppl 1):S25-33. doi: 10.1016/j.ajic.2010.04.196. PMID 20569853
- [Background] Manoukian S, Stewart S, Graves N, Mason H, Robertson C, Kennedy S, Pan J, Haahr L, Dancer SJ, Cook B, Reilly J. Evaluating the post-discharge cost of healthcare-associated infection in NHS Scotland. J Hosp Infect. 2021 Aug;114:51-58. doi: 10.1016/j.jhin.2020.12.026. PMID 34301396
- [Background] Boyce JM. Modern technologies for improving cleaning and disinfection of environmental surfaces in hospitals. Antimicrob Resist Infect Control. 2016 Apr 11;5:10. doi: 10.1186/s13756-016-0111-x. eCollection 2016. PMID 27069623
- [Background] Han JH, Sullivan N, Leas BF, Pegues DA, Kaczmarek JL, Umscheid CA. Cleaning Hospital Room Surfaces to Prevent Health Care-Associated Infections: A Technical Brief. Ann Intern Med. 2015 Oct 20;163(8):598-607. doi: 10.7326/M15-1192. Epub 2015 Aug 11. PMID 26258903
- [Background] Martin ET, Haider S, Palleschi M, Eagle S, Crisostomo DV, Haddox P, Harmon L, Mazur R, Moshos J, Marchaim D, Kaye KS. Bathing hospitalized dependent patients with prepackaged disposable washcloths instead of traditional bath basins: A case-crossover study. Am J Infect Control. 2017 Sep 1;45(9):990-994. doi: 10.1016/j.ajic.2017.03.023. Epub 2017 May 11. PMID 28502637
- [Background] The Israeli Ministry of Health Manual 2006.
- [Background] Marchaim D, Taylor AR, Hayakawa K, Bheemreddy S, Sunkara B, Moshos J, Chopra T, Abreu-Lanfranco O, Martin ET, Pogue JM, Lephart PR, Panda S, Dhar S, Kaye KS. Hospital bath basins are frequently contaminated with multidrug-resistant human pathogens. Am J Infect Control. 2012 Aug;40(6):562-4. doi: 10.1016/j.ajic.2011.07.014. Epub 2011 Dec 16. PMID 22177667
- [Background] Sattar SA, Maillard JY. The crucial role of wiping in decontamination of high-touch environmental surfaces: review of current status and directions for the future. Am J Infect Control. 2013 May;41(5 Suppl):S97-104. doi: 10.1016/j.ajic.2012.10.032. PMID 23622759
- [Background] Baker F, Scott P, Kingsley A. Disposable cleansing wipes. Prof Nurse. 2005 Mar;20(7):45-7. PMID 15754723
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Smith H, Watkins J, Otis M, Hebden JN, Wright MO. Health care-associated infections studies project: An American journal of infection control and national healthcare safety network data quality collaboration case study - Chapter 2 Identifying Healthcare-associated Infections (HAI) for NHSN Surveillance case study vignettes. Am J Infect Control. 2022 Jun;50(6):695-698. doi: 10.1016/j.ajic.2022.02.028. Epub 2022 Mar 8. PMID 35276310
- [Background] Zilberman-Itskovich S, Youngster I, Lazarovitch T, Bondarenco M, Toledano L, Kachlon Y, Mengesha B, Strul N, Zaidenstein R, Marchaim D. Potential impact of removing metronidazole from treatment armamentarium of mild acute Clostridioides difficile infection. Future Microbiol. 2019 Nov;14:1489-1495. doi: 10.2217/fmb-2019-0157. Epub 2020 Jan 8. PMID 31913060
- [Background] Austin PC. Absolute risk reductions and numbers needed to treat can be obtained from adjusted survival models for time-to-event outcomes. J Clin Epidemiol. 2010 Jan;63(1):46-55. doi: 10.1016/j.jclinepi.2009.03.012. Epub 2009 Jul 12. PMID 19595575
- [Background] Tanner WD, Leecaster MK, Zhang Y, Stratford KM, Mayer J, Visnovsky LD, Alhmidi H, Cadnum JL, Jencson AL, Koganti S, Bennett CP, Donskey CJ, Noble-Wang J, Reddy SC, Rose LJ, Watson L, Ide E, Wipperfurth T, Safdar N, Arasim M, Macke C, Roman P, Krein SL, Loc-Carrillo C, Samore MH. Environmental Contamination of Contact Precaution and Non-Contact Precaution Patient Rooms in Six Acute Care Facilities. Clin Infect Dis. 2021 Jan 29;72(Suppl 1):S8-S16. doi: 10.1093/cid/ciaa1602. PMID 33512527
- [Background] Turner RM, White IR, Croudace T; PIP Study Group. Analysis of cluster randomized cross-over trial data: a comparison of methods. Stat Med. 2007 Jan 30;26(2):274-89. doi: 10.1002/sim.2537. PMID 16538700
- [Background] World Health Organization. WHO publishes list of bacteria for which new antibiotics are urgently needed. Published online February 27, 2017
- [Background] Leddin D, Omary MB, Veitch A, Metz G, Amrani N, Aabakken L, Raja Ali RA, Alvares-Da-Silva MR, Armstrong D, Boyacioglu S, Chen Y, Elwakil R, Fock KM, Hamid SS, Makharia G, Macrae F, Malekzadeh R, Mulder CJ, Piscoya A, Perman ML, Sadeghi A, Saenz R, Saurin JC, Butt AS, Wu K, Lee YY. Uniting the Global Gastroenterology Community to Meet the Challenge of Climate Change and Non-Recyclable Waste. Gastroenterology. 2021 Nov;161(5):1354-1360. doi: 10.1053/j.gastro.2021.08.001. Epub 2021 Oct 7. No abstract available. PMID 34629165